CLINICAL TRIAL: NCT00252499
Title: Insulin Resistance in Non-alcoholic Fatty Liver Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol drug change required new clinicaltrails.gov entry
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CDA-2-044-08S
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Results first posted 2014-04-11 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Fatty Liver; Insulin Resistance
Keywords: beta cell function; fenofibrate; non-alcoholic steatohepatitis; rosiglitazone; insulin sensitivity
MeSH Terms: conditions — Fatty Liver; Insulin Resistance; Non-alcoholic Fatty Liver Disease | interventions — Rosiglitazone; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo Arm (Placebo Comparator): matching placebo for rosiglitazone, 1 po bid and placebo for fenofibrate 1 po qd
  Interventions: Drug: placebo for rosiglitazone; Drug: placebo for fenofibrate
- Rosiglitazone Arm (Experimental): rosiglitazone 4 mg po bid and fenofibrate placebo 1 po qd
  Interventions: Drug: rosiglitazone; Drug: placebo for fenofibrate
- Fenofibrate Arm (Experimental): micronized fenofibrate 200 mg 1 po qd and rosiglitazone placebo 1 po bid
  Interventions: Drug: fenofibrate; Drug: placebo for rosiglitazone

INTERVENTIONS:
Drug: rosiglitazone — PPAR-gamma agonist, insulin sensitizer
  Arms: Rosiglitazone Arm
Drug: fenofibrate — PPAR-alpha agonist, reduces triglycerides
  Arms: Fenofibrate Arm
Drug: placebo for rosiglitazone — placebo tablets that are matched to look like rosiglitazone
  Arms: Fenofibrate Arm; Placebo Arm
Drug: placebo for fenofibrate — placebo matched to look like fenofibrate tablets
  Arms: Placebo Arm; Rosiglitazone Arm

SUMMARY:
The purpose of this study is to determine whether nonalcoholic fatty liver disease (NAFLD) is associated with altered peripheral and hepatic insulin sensitivity and to investigate potential mechanisms underlying insulin resistance in NAFLD by determining associations between hepatic and peripheral insulin sensitivity, hepatic steatosis, dyslipidemia, inflammatory cytokines, glucose metabolism, beta-cell function and body fat distribution.

DETAILED DESCRIPTION:
NAFLD and nonalcoholic steatohepatitis (NASH) are common liver disorders that are strongly associated with obesity, type 2 diabetes and dyslipidemia. The underlying pathophysiology of fatty infiltration of the liver is thought to be related to insulin resistance, which is an almost universal finding in patients with NAFLD. It is also possible that fat infiltration and inflammation in the liver may impair insulin sensitivity, either locally in the liver, or peripherally via the actions of inflammatory cytokines. We hypothesize that insulin resistance is a major causal factor leading to fat deposition in the liver and NAFLD, and thus interventions aimed at improving insulin sensitivity will result in a reduction of hepatic inflammation and steatosis.

Specific Aim 1: To determine in a cross-sectional study whether NAFLD is associated with altered peripheral and hepatic insulin sensitivity and to study their relationships with hepatic steatosis, dyslipidemia, inflammatory cytokines, glucose metabolism, -cell function and body fat distribution. Specific Aim 2: To determine in a 6 month placebo-controlled double-blinded treatment study if treatment with rosiglitazone, an insulin sensitizer, or fenofibrate, a triglyceride lowering agent, will improve both hepatic as well as peripheral insulin sensitivity and thereby improve hepatic steatosis and inflammation in subjects with NAFLD.

The results of the proposed study will have important implications for our understanding of the mechanisms underlying insulin resistance and abnormalities in lipid and glucose metabolism in subjects with NAFLD and for the design of future studies aimed at the prevention and treatment of this condition.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old Controls:

  * otherwise healthy Case subjects: NAFLD on liver biopsy within the past 3 years or presumed NAFLD with otherwise unexplained elevated ALT and fatty liver by CT or ultrasound
* Able to comply with taking 3 pills a day for 6 months and follow-up safety visits

Exclusion Criteria:

* Controls:

  * history or evidence of hepatic steatosis
* Cases:

  * Cirrhosis on liver biopsy or by clinical exam or fibrosis score
  * Causes of liver dysfunction other than NASH
* Use of medications associated with hepatic steatosis:

  * glucocorticoids
  * estrogens
  * tamoxifen
  * amiodarone
  * accutane
  * sertraline
* Use of medications that cause insulin resistance:

  * niacin
  * glucocorticoids
  * anti-HIV drugs or atypical antipsychotics
* Use of lipid-lowering medications except stable dose statin
* Use of anti-NASH drugs such as:

  * ursodeoxycholic acid
  * betaine milk thistle
* Use of coumadin
* Use of nitrates
* Significant alcohol consumption:

  * Average >20 grams/day
* In subjects with diabetes

  * a HbA1c >7.5% or use of insulin
  * metformin
  * rosiglitazone or pioglitazone
* Liver transaminases:

  * Cases: ALT >5x upper limit of normal
  * Controls: ALT or AST above the normal range
* Iron saturation >50%
* Creatinine >1.5 mg/dl for men and >1.4 mg/dl for women
* Hematocrit <33%
* Pregnancy or lactation
* Significant weight loss within the past 6 months for controls, or since the liver biopsy for case subjects, history of significant coronary artery disease or congestive heart failure
* Retinopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2005-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Marie Utzschneider, MD, Principal Investigator — VA Puget Sound Health Care System, Seattle
Locations (1):
- VA Puget Sound Health Care System, Seattle, Seattle, Washington, United States

REFERENCES:
- [Result] Utzschneider KM, Largajolli A, Bertoldo A, Marcovina S, Nelson JE, Yeh MM, Kowdley KV, Kahn SE. Serum ferritin is associated with non-alcoholic fatty liver disease and decreased Beta-cell function in non-diabetic men and women. J Diabetes Complications. 2014 Mar-Apr;28(2):177-84. doi: 10.1016/j.jdiacomp.2013.11.007. Epub 2013 Nov 26. PMID 24360972
- [Result] Kratz M, Marcovina S, Nelson JE, Yeh MM, Kowdley KV, Callahan HS, Song X, Di C, Utzschneider KM. Dairy fat intake is associated with glucose tolerance, hepatic and systemic insulin sensitivity, and liver fat but not beta-cell function in humans. Am J Clin Nutr. 2014 Jun;99(6):1385-96. doi: 10.3945/ajcn.113.075457. Epub 2014 Apr 16. PMID 24740208
- See also: Click here for more information about this study: Insulin resistance in non-alcoholic fatty liver disease — http://depts.washington.edu/drgroup/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between 2006 and 2011 through referral from local gastroenterologists.
Pre-assignment Details: Subjects underwent a screening visit prior to randomization to ensure that they qualified for the study.
Groups:
- Arm 1: matching placebo for rosiglitazone, 1 po bid and placebo for fenofibrate 1 po qd
- Arm 2: rosiglitazone 4 mg po bid and fenofibrate placebo 1 po qd
- Arm 3: micronized fenofibrate 200 mg 1 po qd and rosiglitazone placebo 1 po bid
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 5 | 2 | 6
Completed | 4 | 2 | 6
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 5 | 2 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 6 | 13
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (7.3) | 56.5 (4.95) | 54.17 (5.08) | 52.6 (6.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 3 | 1 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Liver/Spleen Ratio at 6 Months
Description: Liver fat was estimated by non-contrast CT scan measuring the density ratio between the liver and spleen by Hounsfield units (liver/spleen ratio), which has been previously correlated with liver fat quantification by magnetic resonance spectroscopy.Ten separate measurements equally distributed throughout the liver and spleen were obtained and the Hounsfield units averaged. In subjects with more than one slice through the liver and spleen, the values for all slices were averaged.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 4 | 2 | 6
ratio | 0.85 (0.08) | 0.96 (0.25) | 0.60 (0.17)

2. Secondary Outcome: Change in Alanine Aminotransferase (ALT) Levels From Baseline to 6 Months
Time Frame: 6 months
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 4 | 2 | 6
U/L | -11.5 (12.9) | -35.0 (37.0) | -15.2 (4.5)

3. Secondary Outcome: Change in the Liver Spleen Ratio by CT Scan From Baseline to 6 Months as a Measure of Fat in the Liver
Time Frame: 6 months
Measure: Mean (Standard Error); unit: ratio
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 4 | 2 | 6
ratio | .09 (.10) | .34 (.09) | -.16 (.10)

4. Secondary Outcome: Change in Peripheral Insulin Sensitivity From Baseline to 6 Months
Description: A two-step stable isotope labeled, hyperinsulinemic-euglycemic clamp procedure was performed with a low dose insulin infusion (20 mU/m2/min) for 3 hours followed by a primed high dose insulin infusion (160 mU/m2/min x 5 minutes then 80 mU/m2/min) for two hours. D20 was infused and adjusted to maintain the blood glucose at 90 mg/dl. Samples for glucose, insulin and 6,6 2d glucose were drawn every 15 minutes during the final half hour of the basal, low dose and high dose insulin periods. Whole body insulin sensitivity was calculated as the rate of glucose disposal (Rd)/lean body mass during the high dose insulin infusion.
Time Frame: 6 months
Population: One person in Arm 1 dropped out and thus is lacking 6 month data. The 6 month isotope data to calculate the rate of glucose disposal was not available for one subject in Arm 3.
Measure: Mean (Standard Error); unit: mg/min/kg
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 4 | 2 | 5
mg/min/kg | 1.65 (2.11) | 0.123 (2.62) | -0.24 (1.14)

5. Secondary Outcome: Changes in Intra-abdominal Fat Area From Baseline to 6 Months
Description: Unenhanced CT scan images were obtained on a General Electric Discovery HD750 CT scanner. Intra-abdominal (IAF) areas were measured at the top of the iliac crest and quantified using the Tomovision program (SliceOMatic V4.3) by one trained technologist.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: mm2
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 5 | 2 | 6
mm2 | 885 (874) | 440 (2788) | 108 (3416)

6. Secondary Outcome: Change in Hepatic Insulin Sensitivity From Baseline to 6 Months
Description: Hepatic insulin sensitivity was determined as the percent suppression of endogenous glucose production (EGP) at the end of the low dose insulin clamp.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: percent of baseline EGP
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 4 | 2 | 5
percent of baseline EGP | 23.3 (7.8) | -4.09 (4.34) | 4.91 (9.32)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2 | Arm 3
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 3/5 | 0/2 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=5) | Arm 2 (N=2) | Arm 3 (N=6)
gout attack (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (3)
vasovagal reaction (General disorders) | 2 (2) | 0 (0) | 0 (0)
leg edema (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
increased serum Creatinine (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Due to recruitment difficulties and concerns about the safety of thiazolidinediones, recruitment was stopped without achieving adequate sample size (16/arm). Thus, no definitive conclusions can be made about the study medications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes